CLINICAL TRIAL: NCT04253327
Title: Impact of Diagnosis and Surgical Treatment of Borderline Ovarian Tumors on Distress, Anxiety and Psychosexual Health
Brief Title: Distress, Anxiety and Psychosexual Health in BOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Stefan Cosyns, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: sBOT D/A/PSH
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Ovarian Neoplasm Epithelial Borderline
Keywords: low malignant potential; sexual health; anxiety; distress; surgery
MeSH Terms: conditions — Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BOT: Patients diagnosed and treated by surgery for borderline ovarian tumor
  Interventions: Other: questionnaire
- controls: Patients after surgical treatment of benign ovarian tumor
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Patients will be contacted by their physician during regular follow-up in the out-patient clinic or contacted by phone.
  The questionnaires will be filled in at the UZBrussel, Laarbeeklaan 101, 1090 Brussels or at the patients home.
  Filled-in questionnaires can be hand off immediately at the physician or send by post or email..

SUMMARY:
The aim of this study is to assess the prevalence of distress, anxiety and psychosexual anguish in patients diagnosed with borderline ovarian tumor (BOT) compared to controls confronted with surgical treatment for benign ovarian tumors.

DETAILED DESCRIPTION:
Appropriate surgical care is primordial for the patient after diagnosis of a BOT. Taking into account the good prognosis and long live expectancy caregivers should also be concerned about non-oncological complains during the follow-up to guarantee the overall well-being of the patient.

Women diagnosed with gynaecological cancer are likely to face additional consequences beyond those common to all cancer patients.

Not surprisingly, previous research shows that women affected by gynaecological cancer are likely to suffer significant physical and psychological morbidity. Studies including women of all ages with gynaecological cancers indicate higher levels of psychological distress, including clinical levels of anxiety, depression and posttraumatic distress disorder as well as greater decrements in body image and more sexual problems than in other types of cancer. High levels of distress were reported up to four years following the diagnosis.

Longitudinal studies addressing the prevalence of psychological distress, anxiety or psychosexual health during follow up in BOT patients are lacking. Due to the connotation between sexuality and internal genitals, diagnosis of the BOT and following surgery are possibly negatively influencing each other. Large prospective or randomized control studies are unachievable due to the low prevalence of BOT and limited recurrences or death.

Identification of the presence of psychological morbidity, including anxiety and depression is clinically useful because, unlike most demographic and clinical factors, psychological illness and psychosexual complaints are modifiable.

The study material consists out of two main parts of questionnaires.

A first questionnaire addressing the distress and anxiety consists of validated questionnaires:

* Hospital Anxiety and Depression Scale (HADS),
* Body Image Scale (BIS),
* Perceived Stress Scale (PSS).

And a second questionnaire concerning psychosexual health, built up out of validated questionnaires;

* Female Sexual Function Index (FSFI),
* Female Sexual Distress Scale - Revised (FSDS-R),
* European Organisation for Research and Treatment of Cancer (EORTC) quality of life (QOL) questionnaire designed to measure the QOL of patients with ovarian cancer (EORTC QLQ-OV28) (only questions 50-58)
* EORTC Sexual Health Questionnaire (EORTC SHQ-C22) for assessing sexual health in cancer patients (only the part concerning women).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis and surgery for benign or borderline ovarian tumors.
* >18 y.

Exclusion Criteria:

* Known former psychological morbidity evaluated by the investigators.
* History of another cancer type.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having had surgery for benign or borderline ovarian tumors
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety and Depression - HADS | 2020
  Anxiety and depression will be measured using a validated questionnaire: Hospital Anxiety and Depression Scale - The scores for anxiety and depression can vary from 0 to 21, depending on the presence and severity of the symptoms. A score between 0 and 7 does not indicate the presence of the symptoms; a score between 8 and 10 indicates the presence of the symptoms but to a moderate degree, therefore doubtful cases; a score greater than or equal to 11 indicates a significant number of symptoms corresponding to confirmed cases.
Depression - BIS | 2020
  Depression will be measured using two validated questionnaires. The first one will be the Body Image Scale (BIS). The BIS is a a 10-item scale informing about self-image. A low score is reflecting a low body image.
Anxiety - Perceived Stress Scale | 2020
  The validated questionnaire measuring perceived stress among our study population will be the Perceived Stress Scale or PSS.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Psycho-sexual health - FSFI | 2020
  Psychosexual health will be measured using different validated questionnaires: The First will be the Female sexual function index (FSFI). This is a 19-item questionnaire provides scores on six domains of sexual function (desire, arousal, lubrication, orgasm, satisfaction, and pain) as well as a total score. A score ≤ 26.55 is classified as a Female Sexual Disorder.
Psycho-sexual health - FSDS - Revised | 2020
  Psycho-sexual health will be measured using different validated questionnaires: As second we will use is the Female sexual distress scale (FSDS-R), a 13-item questionnaire designed to measure sexually related personal distress in women. A low score reflects a normal sexual health whereas a high score an in-satisfaction about the sexual health reflects.
Psycho-sexual health - EORTC OV28 | 2020
  Psychosexual health will be measured using different validated questionnaires: The third questionnaire is one of the EORTC quality of life questionnaire for patient with ovarian cancer (EORTC QLQ-OV28). The EORTC QLQ questionnaire is designed to measure quality of life in cancer patients. A high score for the [functional scales and/or single items] represents a high level of functioning, whereas a high score for the [symptom scales and/or single items] represents a high level of symptomatology or problems.
Psycho-sexual health - EORTC SHQ C22 | 2020
  Psycho-sexual health will be measured using different validated questionnaires: The last questionnaire will be the EORTC Sexual health questionnaire for cancer patients (EORTC SHQ-C22). This questionnaires is designed to measure sexual health in cancer patients. A high score for the [functional scales and/or single items] represents a high level of functioning, whereas a high score for the [symptom scales and/or single items] represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis UZBrussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cosyns S, Dony N, Polyzos N, Buyl R, Tournaye H, Schotte C. Impact of diagnosis and surgical treatment of early stage borderline ovarian tumours on distress, anxiety, and psychosexual health. J Psychosom Obstet Gynaecol. 2024 Dec;45(1):2404010. doi: 10.1080/0167482X.2024.2404010. Epub 2024 Sep 20. PMID 39301872